CLINICAL TRIAL: NCT02426775
Title: Randomized Multicentre Comparative Trial to Evaluate the Long Term Effectiveness of the Use of Carbaglu® in Patients With Propionic Acidemia (PA) or Methylmalonic Acidemia (MMA)
Brief Title: Carglumic Acid in Methylmalonic Acidemia and Propionic Acidemia
Acronym: CAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Dr. Majid Alfadhel, Head Genetics Division, Department of Pediatrics. Assistant Professor, King Saud bin Abdulaziz University for Health Sciences (KSAU-HS), King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 13/116
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Propionic Acidemia; Methylmalonic Acidemia
MeSH Terms: conditions — Propionic Acidemia; Methylmalonic acidemia | interventions — carglumic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methylmalonic Acidemia Control Arm (No Intervention): patients with Methylmalonic Acidemia will receive standard therapy only (protein restricted diet, L-carnitine, metronidazole and vitamin B12)
- Methylmalonic Acidemia Active arm (Experimental): patients with Methylmalonic Acidemia will receive Carglumic Acid in addition to standard therapy (protein restricted diet, L-carnitine, metronidazole and vitamin B12)
  Interventions: Drug: Carglumic Acid
- Propionic Acidemia Control Arm (No Intervention): patients with Propionic Acidemia will receive standard therapy only (protein restricted diet, L-carnitine, metronidazole and biotin)
- Propionic Acidemia Active arm (Experimental): patients with Propionic Acidemia will receive Carglumic Acid in addition to standard therapy (protein restricted diet, L-carnitine, metronidazole and biotin)
  Interventions: Drug: Carglumic Acid

INTERVENTIONS:
Drug: Carglumic Acid — Carglumic Acid 50 mg/kg/day (twice daily)
  Other Names: Carbaglu
  Arms: Methylmalonic Acidemia Active arm; Propionic Acidemia Active arm

SUMMARY:
A Phase IIIb (Three b), Randomized Multicentre Comparative Trial to Evaluate the Long Term Effectiveness & Safety of the use of Carglumic Acid (Carbaglu®) in Patients with Propionic Acidemia (PA) or Methylmalonic Acidemia (MMA). Carbaglu® clinical experience in Organic Acidemia (OA) is limited to a non-comparative retrospective collection of data from patients who had received Carbaglu® for 1 to 15 days.

There is no current evidence supporting the use of carglumic acid for the chronic management of patients with OA. The investigators are proposing a randomized multicentre prospective clinical trial to evaluate long-term effects of the use of Carbaglu® (50mg/kg/day) combined with standard chronic therapy in patients with PA and MMA compared to standard chronic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Children of 15 years old or less
* Parent or legal guardian agree to participate and to sign the (Institutional Review Board) IRB approved Informed Consent Form (assent forms will be waived due to the mental disability of those children)
* Not participating in any other clinical trial in the previous 30 days
* PA or MMA confirmed using the following criteria:

  * PA confirmed by the measurement of acylcarnitine profile, urine organic acid, measurement of propionyl Co-A carboxylase in leukocytes or cultured fibroblasts or by DNA molecular testing of PCCA (Propionyl CoA Carboxylase, Alpha Polypeptide) or PCCB (propionyl CoA carboxylase, beta polypeptide) gene
  * MMA confirmed by the measurement of acylcarnitine profile, urine organic acid, measurement of methymalonyl Co-A mutase in culture fibroblasts or DNA molecular testing of mutgene.
* Expected survival of at least 6 months, for the purpose of this study Survival expectance will be defined as patient not admitted to the Pediatric Intensive Care Unit (PICU) due to hyperammonemia more than 2 times per year or asymptomatic patients diagnosed by newborn screening program or stable chronic patients who are followed up at outpatient clinic.

Exclusion Criteria:

* Patients with other organic acidemia or any other cause of hyperammonemia
* Patient receiving other investigational therapy for PA or MMA
* Past history of hypersensitivity or drug allergy to Carbaglu®
* Patient with PA or MMA and other inherited genetic conditions or congenital anomalies

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Number of emergency visits due to hyperammonemia within 24 months period | 24 months

SECONDARY OUTCOMES:
Time to first visit to the ER due to hyperammonemia from starting the treatment. | 24 months
Plasma ammonia levels over the study treatment period. | 24 months
Number of days of hospitalization | 24 months
Acylcarnitine level for all patients | once on screening visit
Measuring urine organic acid levels for both diseases. | 24 months
Measuring Plasma aminoacids' levels for both diseases | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Majid A. Alfadhel, MD, Principal Investigator — King Abdulaziz Medical City, National Guard / Riyadh-Saudi Arabia
Locations (2):
- Saudi Arabia (2):
  - King Abdullah Specialist Children Hospital, King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh

REFERENCES:
- [Derived] Nashabat M, Obaid A, Al Mutairi F, Saleh M, Elamin M, Ahmed H, Ababneh F, Eyaid W, Alswaid A, Alohali L, Faqeih E, Aljeraisy M, Hussein MA, Alasmari A, Alfadhel M. Evaluation of long-term effectiveness of the use of carglumic acid in patients with propionic acidemia (PA) or methylmalonic acidemia (MMA): study protocol for a randomized controlled trial. BMC Pediatr. 2019 Jun 13;19(1):195. doi: 10.1186/s12887-019-1571-y. PMID 31196016